CLINICAL TRIAL: NCT06923319
Title: Learning Curves for Odòn, Kiwi Vacuum, and Simpson Forceps for Vaginal Birth on Mannequin
Brief Title: Learning Curves of Different Devices for Vaginal Birth on Mannequin
Status: Enrolling by invitation | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Claudio Celentano, Head of Unit, G. d'Annunzio University
Other Study IDs: ObGynEASC008
Record Dates: First submitted 2025-03-21; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Forceps Delivery Affecting Fetus or Newborn; Ventouse Extraction;Liveborn; Birth; Forced
Keywords: Odòn; Kiwi vacuum; Simpson forceps

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Odòn device: learning time 0, 1 month and 2 month
  Interventions: Device: Odòn, Kiwi, Simpson skills
- Kiwi vacuum: learning time 0, 1 month and 2 month
  Interventions: Device: Odòn, Kiwi, Simpson skills
- Simpsong forceps: learning time 0, 1 month and 2 month
  Interventions: Device: Odòn, Kiwi, Simpson skills

INTERVENTIONS:
Device: Odòn, Kiwi, Simpson skills — time 0, time 1 month and 2 months
  Other Names: retaining of skills

SUMMARY:
Learning curves for residents and specialists for devices applied on operative vaginal birth on mannequin (Odòn, Kiwi, Simpson forceps)

DETAILED DESCRIPTION:
Residents and specialists were exposed to formal lecture having the opportunity of digital evaluation of digital support. After a frontal lecture they will have a formal explanation of mannequin approach for each device (Odòn, Kiwi, Simpson) After one month and after two month they will re-train on mannequin for each device.

Before frontal lecture they will answer to a questionnaire evaluating status of residency (year), elderly of specialization (years after degree) and personal experience in labor ward and on mannequin for training. After each training session they will have a further questionnaire evaluating how the training was working on their knowledge and on retaining of skills.

All training sessions will be recorded in a blind way erasing voice and face and with a ID computer generated code.

All videos will be evaluated by three different specialists of known experience on the three devices

ELIGIBILITY:
Inclusion Criteria:

* residents
* specialists

Exclusion Criteria:

* none

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ObGyn specialists and residents involved on Labor ward in Pescara Hospital (above 2000 deliveries per year)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Learning curve | time 0
  rate of success for each device on mannequin
retaining of skills | time 1 month
  rate of success for each device on mannequin
retaining of skills | time 2 months
  rate of success for each device on mannequin

SECONDARY OUTCOMES:
physician approach | time 0, 1 onth and 2 months
  subjective approach to the device
residency and year of specialist approach | time 0, 1 month, and 2 months
  previous experience and clinical status of trainers

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University of Chieti, Chieti, CH
  - Santo Spirito Hospital, Pescara, PE

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet